CLINICAL TRIAL: NCT04715659
Title: A Novel Incremental Step Test as an Alternative for the Assessment of Exercise Capacity in Patients With COPD - The Study of Its Measurement Properties
Brief Title: A Novel Incremental Step Test as an Alternative for the Assessment of Exercise Capacity in Patients With COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Polytechnic Institute of Porto (Other)
Collaborators: Nippon Gases Portugal (Unknown)
Responsible Party: Principal Investigator, Rui Vilarinho, Professor, Polytechnic Institute of Porto
Other Study IDs: reabilitar_DPOC
Record Dates: First submitted 2021-01-03; First posted 2021-01-20 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: COPD
Keywords: validity; reliability; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients
  Interventions: Diagnostic Test: Performance of step test (number of steps) for the assessment of exercise capacity

INTERVENTIONS:
Diagnostic Test: Performance of step test (number of steps) for the assessment of exercise capacity — The development of the step test will be designed according to the characteristics of other validated field tests - the walking tests (6-minute walk test and the incremental shuttle walking test) The step test will be performed on a 20 cm tall, single-step device with no handles. The criteria for stopping the test will be the same as described in standard operating procedures for the walking field tests, with the addition of the inability to follow the work rate for a period of 10 seconds.
  The main outcome of the test will be the highest number of steps and work rate achieved.

SUMMARY:
According to the official guidelines of pulmonary rehabilitation, a structured home-based approach is recommended to answer to the inadequate number of pulmonary rehabilitation services due to the chronic obstructive pulmonary disease (COPD) patient's needs. For this new setting, new strategies for the assessment of exercise capacity and exercise training are essential. The modality of step can be a promising tool because it is inexpensive, portable, and reflects one of the main activities of daily living (stair climbing). The development of a new field test implies the study of the measurement properties, to facilitate the selection of tests and the interpretation of the results in rehabilitation. This project hypothesizes that the step test can be valid, reliable, and feasible to apply in this new setting of pulmonary rehabilitation.

DETAILED DESCRIPTION:
The primary aim of this project is to develop and determine the measurement properties (validity and reliability) of a novel step test for the assessment of exercise capacity in patients with COPD.

The investigators will perform two cross-sectional studies for validity and reliability in patients with COPD. Participants attending a pneumology consultation at the hospital will be asked for permission to be contacted about the study. The participants who agree will be seen by the principal investigator who will explain the nature of the study and assess eligibility for the study. The participants will sign informed consent.

The validity study will be performed in two days (separated >48h). During the first session, the participants will perform the 6-minute walk test (6MWT) twice (a valid test for COPD). On the second day, the step test will be performed twice.

The reliability study will be performed in two days (separated for 7 days). On both days, the step test will be performed one time.

The investigators predict that 50 patients with COPD will be followed in each study (validity and reliability).

The investigators hypothesize that the step test can be a good option to apply in pulmonary rehabilitation programs with good measurement properties for the assessment of exercise capacity in COPD patients. The validation of the test can contribute to applying the step modality in the exercise training as an alternative for the prescription of the exercise intensity. For that, the investigators also hypothesize that the test can be reliable and one test must be enough for the assessment of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible with a diagnose of chronic obstructive pulmonary disease (COPD).

Exclusion Criteria:

* Patients will be excluded if they have a significant cardiac, immune, musculoskeletal or neurological impairment, or any other that does not allow them to perform the tests.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending a pneumology consultation at the hospital will be asked for permission to be contacted about the study. Those who agree will be seen by the principal investigator who will explain the nature of the study and assess eligibility for the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of steps | Through test completion, duration of the test 15 minutes
  The primary outcome will be the amount of the number of steps performed in the step test
Distance walked | Through test completion, duration of the test 6 minutes
  The primary outcome will be the distance walked performed in the 6-minute walk test
Distance walked | Through test completion, duration of the test 12 minutes
  The primary outcome will be the distance walked performed in the incremental shuttle walk test

SECONDARY OUTCOMES:
Dyspnea during the tests | Through test completion, duration of the tests 6 and 15 minutes
  Dyspnea experienced during the tests, monitored with the modified Borg scale, that ranges from 0 to 10, where 0 represents no dyspnea and 10 the worst dyspnea.
Fatigue during the tests | Through test completion, duration of the tests 6 and 15 minutes
  Fatigue experienced during the tests, monitored with the modified Borg scale, that ranges from 0 to 10, where 0 represents no fatigue and 10 the worst fatigue
Heart rate during the tests | Through test completion, duration of the tests 6 and 15 minutes
  Heart rate assessed during the tests, monitored with a cardiofrequencimeter
Oxygen saturation during the tests | Through test completion, duration of the tests 6 and 15 minutes
  Oxygen saturation assessed during the tests, monitored with a pulse oximeter

CONTACTS AND LOCATIONS:
Locations (1):
- Rui Vilarinho, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goncalves T, Carlos Winck J, Silva F, Caneiras C, Montes AM, Vilarinho R. Measurement properties of the incremental step test for people with chronic obstructive pulmonary disease: a cross-sectional study. BMJ Open. 2024 Feb 7;14(2):e078425. doi: 10.1136/bmjopen-2023-078425. PMID 38326260
- [Derived] Vilarinho R, Serra L, Aguas A, Alves C, Silva PM, Caneiras C, Montes AM. Validity and reliability of a new incremental step test for people with chronic obstructive pulmonary disease. BMJ Open Respir Res. 2022 Apr;9(1):e001158. doi: 10.1136/bmjresp-2021-001158. PMID 35387847